Official Title: An Open-Label, Single-Arm, Phase 1/2 Study Evaluating the Safety and Efficacy of Itacitinib in Participants With Bronchiolitis Obliterans Syndrome Following Lung Transplantation

NCT Number: NCT03978637

Document Date: Statistical Analysis Plan Amendment Version 1: 26 August 2024

# **Statistical Analysis Plan**



### INCB 39110-214

# An Open-Label, Single-Arm, Phase 1/2 Study Evaluating the Safety and Efficacy of Itacitinib in Participants With Bronchiolitis Obliterans Syndrome Following Lung Transplantation

| IND Number: | 109,296 |
|---|---|
| <b>EudraCT Number:</b> | 2019-004171-39 |
| Sponsor: | Incyte Corporation<br>1801 Augustine Cut-Off<br>Wilmington, DE 19803 |
| <b>Protocol Version:</b> | Protocol Amendment (Version 3) dated 11 AUG 2020 |
| <b>CRF Approval Date:</b> | 22 SEP 2020 |
| SAP Version: | Amendment 1 |
| SAP Author: | , PhD , Biostatistics |
| Date of Plan: | 26 AUG 2024 |

This study is being conducted in compliance with Good Clinical Practice, including the archiving of essential documents.

# **TABLE OF CONTENTS**

| TITLE PAG | GE | 1 |
|-----------|-----------------------------------------------------------|----|
| TABLE OF | F CONTENTS | 2 |
| LIST OF A | BBREVIATIONS | 5 |
| 1. | INTRODUCTION | 7 |
| 2. | STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS | 8 |
| 2.1. | Protocol and Case Report Form Version | 8 |
| 2.2. | Study Objectives and Endpoints | 8 |
| 3. | STUDY DESIGN | 10 |
| 3.1. | Randomization | 10 |
| 3.2. | Control of Type I Error | 10 |
| 3.3. | Sample Size Considerations | 11 |
| 3.4. | Schedule of Assessments | 11 |
| 4. | DATA HANDLING DEFINITIONS AND CONVENTIONS | 11 |
| 4.1. | Scheduled Study Evaluations and Study Periods | 11 |
| 4.1.1. | Day 1 | 11 |
| 4.1.2. | Study Day | 11 |
| 4.1.3. | Baseline Value | 11 |
| 4.1.4. | Last Available Value | 11 |
| 4.1.5. | Handling of Missing and Incomplete Data | 12 |
| 4.2. | Variable Definitions. | 12 |
| 4.2.1. | Body Mass Index | 12 |
| 4.2.2. | Prior and Concomitant Medication | 12 |
| 4.2.3. | Creatinine Clearance | 12 |
| 5. | STATISTICAL METHODOLOGY | 13 |
| 5.1. | General Methodology | 13 |
| 5.2. | Treatment Groups | 13 |
| 5.3. | Analysis Populations | 13 |
| 5.3.1. | Full Analysis Set. | 13 |
| 5.3.2. | Pharmacokinetic-Evaluable Population | 13 |
| 6. | BASELINE, EXPOSURE, AND DISPOSITION | 14 |
| 6.1 | Demographics Baseline Characteristics and Medical History | 14 |

| 6.1.1. | Demographics and Baseline Characteristics | 14 |
|---|---|---|
| 6.1.2. | Medical History | 14 |
| 6.1.3. | Lung Transplant History | 14 |
| 6.1.4. | Bronchiolitis Obliterans Syndrome History | 14 |
| 6.1.5. | Medications for Immunosuppression | 14 |
| 6.1.6. | Medications for Treatment of Bronchiolitis Obliterans Syndrome | 15 |
| 6.2. | Disposition of Participants | 15 |
| 6.3. | Protocol Deviations | 15 |
| 6.4. | Exposure | 15 |
| 6.5. | Study Drug Compliance | 15 |
| 6.6. | Prior and Concomitant Medication | 15 |
| 7. | EFFICACY | 16 |
| 7.1. | General Considerations | 16 |
| 7.2. | Efficacy Hypotheses | 16 |
| 7.3. | Analysis of the Primary Efficacy Parameter | 16 |
| 7.4. | Analysis of the Secondary Efficacy Parameter | 16 |
| 7.4.1. | Duration of FEV <sub>1</sub> Response | 16 |
| 7.4.2. | Time to Progression or Death | 17 |
| 7.4.3. | SGRQ Total Score | 17 |
| 7.4.4. | QOL-SF-12 Questionnaire | 17 |
| 7.4.5. | EQ-5D-3L | 18 |
| 8. | PHARMACOKINETICS AND PHARMACODYNAMICS | 19 |
| 8.1. | Pharmacokinetic Analyses | 19 |
| 8.1.1. | Pharmacokinetic Data | 19 |
| 8.1.2. | Participant Demographic, Clinical Laboratory, Disease-Related, and Pharmacogenomic Variables and Concomitant Medications | 19 |
| 8.1.3. | Pharmacokinetic Analyses | 19 |
| 8.1.4. | Report | 20 |
| 8.2. | Pharmacodynamic Analyses | 20 |
| 9. | SAFETY AND TOLERABILITY | 21 |
| 9.1. | General Considerations | 21 |
| 9.2. | Adverse Events | 21 |
| 9.2.1. | Adverse Event Definitions | 21 |

### LIST OF FIGURES

# LIST OF ABBREVIATIONS

| Abbreviation | Term |
|---|---|
| AE | adverse event |
| AUC <sub>0-t</sub> | area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t |
| AUC <sub>0-τ</sub> | area under the steady-state plasma or serum concentration-time curve over 1 dose interval |
| BMI | body mass index |
| BOS | bronchiolitis obliterans syndrome |
| CI | confidence interval |
| Cl/F | apparent oral dose clearance |
| C <sub>max</sub> | maximum observed plasma or serum concentration |
| C <sub>min</sub> | minimum observed plasma or serum concentration over the dose interval |
| CMV | cytomegalovirus |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| EBV | Epstein-Barr virus |
| ECP | extracorporeal photopheresis |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOT | end of treatment |
| EQ-5D-3L | EuroQol 5-dimension 3-level |
| EQ-VAS | EuroQol visual analogue scale |
| EU | European Union |
| FAS | full analysis set |
| FEV <sub>1</sub> | forced expiratory volume in 1 second |
| FDA | Food and Drug Administration |
| GVHD | graft-versus-host disease |
| HDL | high-density lipoprotein |
| JAK | Janus kinase |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI | National Cancer Institute |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| QOL-SF-12 | Quality of Life 12-Item Short Form |
| QOL-SF-36 | Quality of Life 36-Item Short Form |
| QTcB | QT interval corrected using Bazett's formula |
| QTcF | QT interval corrected using Fridericia's formula |
| RP2D | recommended Phase 2 dose |

| Abbreviation | Term |
|-------------------|--------------------------------------------------|
| SAP | Statistical Analysis Plan |
| SGRQ | St George's Respiratory Questionnaire |
| SOC | system organ class |
| STAT | signal transducer and activator of transcription |
| t <sub>1/2</sub> | half-life |
| TEAE | treatment-emergent adverse event |
| t <sub>max</sub> | time to maximum concentration |
| US | United States |
| V <sub>z</sub> /F | apparent oral dose volume of distribution |
| WHO | World Health Organization |

#### 1. INTRODUCTION

Post—lung transplant BOS is a serious, life-threatening condition which represents a significant unmet medical need. There are few therapeutic trials for BOS, and currently no agents are approved by the FDA for the treatment of BOS. Treatments used in clinical practice are associated with significant toxicities and high failure rates.

Novel treatments with agents targeting JAK-STAT pathways appear to decrease alloreactive T-cell damage in both preclinical models of GVHD as well as in completed and ongoing clinical trials. The biology of GVHD shares many similar mechanisms with post–lung transplant BOS and it is hypothesized that the selective JAK1 inhibitor, itacitinib, may be an effective therapy for post–lung transplant BOS.

Study INCB 39110-214 is a Phase 1/2 study that will evaluate itacitinib in post–lung transplant Grade 1 through 3 BOS. The study design comprises a randomized, open-label, parallel dose selection run-in followed by a single arm expansion to evaluate the efficacy in this population.

The purpose of this SAP is to provide details of the statistical analyses that have been outlined in the Protocol.

### 2. STUDY INFORMATION, OBJECTIVES, AND ENDPOINTS

# 2.1. Protocol and Case Report Form Version

This SAP is based on INCB 39110-214 Protocol Amendment (Version 3) dated 11 AUG 2020 and CRFs approved 22 SEP 2020. Unless superseded by an amendment, this SAP will be effective for all subsequent Protocol amendments and eCRF versions.

### 2.2. Study Objectives and Endpoints

Table 1 presents the objectives and endpoints.

**Table 1:** Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| Phase 1 | |
| To identify an appropriate dose of itacitinib as a treatment for Grade 1 through 3 BOS following lung transplantation. | Frequency, severity, and duration of AEs; assessment of changes in safety and FEV <sub>1</sub> ; and assessment of changes in laboratory parameters, PK, and pharmacodynamics. |
| Phase 2 | |
| To evaluate the efficacy of itacitinib as a treatment for Grade 1 through 3 BOS following lung transplantation. | FEV <sub>1</sub> response rate from baseline through the Week 12 visit, defined as the proportion of participants demonstrating a $\geq$ 10% absolute increase in FEV <sub>1</sub> compared to baseline. |
| Secondary | |
| Phase 1 and Phase 2 | |
| To evaluate duration of FEV <sub>1</sub> response in participants with Grade 1 through 3 BOS following lung transplantation who are treated with itacitinib. | Duration of FEV <sub>1</sub> response, defined as the time of the onset of response ( $\geq 10\%$ absolute increase in FEV <sub>1</sub> compared to baseline) to BOS progression ( $\geq 10\%$ absolute decrease in FEV <sub>1</sub> compared to baseline) or loss of clinical benefit as determined by the investigator. |
| To evaluate time to progression in participants with Grade 1 through 3 BOS following lung transplantation who are treated with itacitinib. | Time to progression, defined as the interval between the start of treatment and BOS progression (≥ 10% absolute decrease in FEV₁ compared to baseline), or death. |
| To evaluate quality of life outcomes in participants with Grade 1 through 3 BOS following lung transplantation who are treated with itacitinib. | <ul> <li>Change from baseline in SGRQ total score.</li> <li>Change from baseline in QOL-SF-12 questionnaire.</li> <li>Categorical summary or change from baseline in EQ-5D-3L questionnaire.</li> </ul> |
| To evaluate the PK of itacitinib in the study population. | C <sub>max</sub> , C <sub>min</sub> , t <sub>max</sub> , AUC <sub>0-t</sub> , and Cl/F. |

**Table 1:** Objectives and Endpoints (Continued)

| Objectives | Endpoints |
|---|---|
| Secondary (continued) | |
| Phase 2 only | |
| To evaluate overall survival or time to retransplantation in participants with Grade 1 through 3 BOS following lung transplantation who are treated with itacitinib. | Time to retransplantation or death, defined as the interval between the start of treatment and the date of retransplantation or death due to any cause. |

#### 3. STUDY DESIGN

This Phase 1/2 study will evaluate the safety, efficacy, PK, and pharmacodynamics of itacitinib in participants with post–lung transplant BOS.

Phase 1 is a dose selection run-in that will employ a randomized, open-label, parallel-cohort design to assess the safety, tolerability, PK, and pharmacodynamics and determine the RP2D of itacitinib in participants with post–lung transplant BOS. A total of 24 participants with Grade 1, 2, or 3 BOS will be assigned to receive 1 of 3 itacitinib dose levels (n = 8 each). Each Phase 1 dose level will enroll a maximum of 2 participants with Grade 3 BOS. Participants will be randomized to 1 of 3 dose levels using an interactive response technology system. Upon completion of Phase 1 enrollment, the RP2D will be selected on the basis of AE, laboratory, PK, and pharmacodynamic observations through the Week 12 visit. Additionally, an efficacy analysis will be performed to determine the FEV<sub>1</sub> response rate for all participants treated for  $\geq$  12 weeks. The study will proceed to Phase 2 if  $\geq$  1 responses (defined as  $\geq$  10% absolute increase in FEV<sub>1</sub> compared with baseline, confirmed by 2 consecutive spirometric assessments  $\geq$  1 week apart) are observed at the dose level selected as the RP2D.

Phase 2 will employ a single-arm, open-label design to evaluate the efficacy and further characterize the safety of itacitinib at the RP2D.

Itacitinib treatment in Phase 1 and Phase 2 will continue until progression of BOS (defined as a  $\geq 10\%$  absolute decrease from baseline in FEV<sub>1</sub>, confirmed by 2 consecutive spirometric assessments  $\geq 3$  weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.

Figure 1 presents the study design schema.

Figure 1: Study Design Schema



<sup>&</sup>lt;sup>a</sup> Not inclusive.

#### 3.1. Randomization

In Phase 1, approximately 24 participants will be randomly assigned to receive 1 of 3 itacitinib dose levels in a 1:1:1 allocation ratio.

# 3.2. Control of Type I Error

No formal efficacy hypotheses will be tested, and no alpha control will be implemented.

### 3.3. Sample Size Considerations

In Phase 1, approximately 24 participants will be enrolled to participate across the 3 dose levels of itacitinib to identify the RP2D. A sample size of 24 participants (8 per dose level) allows for concurrent enrollment at 3 dose levels that have been previously characterized in other disease settings and is expected to enable the clinical characterization of safety and efficacy.

In Phase 2, the FEV<sub>1</sub> response rate for itacitinib is assumed to be 20%. In order for the lower confidence limit of the 95% CI to exclude 5%, approximately 55 participants are needed.

#### 3.4. Schedule of Assessments

Refer to Protocol Amendment (Version 3) dated 11 AUG 2020 for a full description of all study procedures and assessment schedules for this study.

#### 4. DATA HANDLING DEFINITIONS AND CONVENTIONS

### 4.1. Scheduled Study Evaluations and Study Periods

#### 4.1.1. Day 1

Day 1 is the date the first dose of itacitinib is administered to the participants.

### **4.1.2. Study Day**

If a visit/reporting date is on or after Day 1, then the study day at the visit/reporting date will be calculated as

```
Day \# = (visit/reporting date - Day 1 date + 1)
```

If the visit/reporting date is before Day 1, then the study day at the visit/reporting date will be calculated as

```
Day # = (visit/reporting date - Day 1 date)
```

A study day of -1 indicates 1 day before Day 1.

#### 4.1.3. Baseline Value

Baseline is the last nonmissing measurement obtained before the first administration of itacitinib.

When scheduled assessments and unscheduled assessments occur on the same day, and time of the assessment or time of first dose is not available, use the following convention to determine baseline: if both a scheduled and an unscheduled visit are available, use the scheduled assessment as baseline.

#### 4.1.4. Last Available Value

The last available value is the last nonmissing measurement obtained after starting itacitinib.

#### 4.1.5. Handling of Missing and Incomplete Data

In general, values for missing data will not be imputed unless methods for handling missing data are specified in this section or relevant sections.

#### 4.2. Variable Definitions

#### 4.2.1. Body Mass Index

Body mass index will be calculated as follows:

BMI  $(kg/m^2) = [weight (kg)] / [height (m)]^2$ 

#### 4.2.2. Prior and Concomitant Medication

Prior medication is defined as any nonstudy medication started and stopped before the first dose of itacitinib.

Concomitant medication is defined as any nonstudy medication that is started accordingly:

- Before the date of first administration of itacitinib and is ongoing throughout the study or ends on/after the date of first administration of itacitinib.
- On/after the date of first administration of itacitinib and is ongoing or ends during the course of the study.

A prior medication could also be classified as "both prior and concomitant medication" if the end date is on or after first dose of itacitinib. In the listing, it will be indicated whether a medication is prior-only, concomitant-only, or both prior and concomitant.

For the purposes of analysis, all medications will be considered concomitant medications unless the medications can unequivocally be defined as not concomitant.

#### 4.2.3. Creatinine Clearance

Creatinine clearance by Cockcroft-Gault equation (Cockcroft and Gault 1976) is estimated from serum creatinine (mg/dL) determination using the following formula:

Creatinine clearance (mL/min) =  $[140 - age (years)] \times weight (kg) \times \{0.85 \text{ for female participants}\} / [72 \times serum creatinine (mg/dL)]$ 

#### 5. STATISTICAL METHODOLOGY

### **5.1.** General Methodology

Unless otherwise noted, SAS® software (SAS Institute Inc, Cary, NC; v9.4 or later) will be used for the generation of all tables, graphs, and statistical analyses. Descriptive summaries for continuous variables will include, but not be limited to, the number of observations, mean, standard deviation, median, minimum, and maximum. Descriptive summaries for categorical variables will include the number and percentage of participants in each category.

### **5.2.** Treatment Groups

In Phase 1, a total of 24 participants with Grade 1, 2, or 3 BOS will be assigned to receive 1 of 3 itacitinib dose levels (n = 8 each).

In Phase 2, participants will be treated with itacitinib at the RP2D.

### 5.3. Analysis Populations

#### 5.3.1. Full Analysis Set

The FAS will include all participants enrolled in the study who received at least 1 dose of itacitinib. The FAS will be used for the summary of demographics, baseline characteristics, participant disposition, and analyses of all safety, study treatment administration, and efficacy data.

### **5.3.2.** Pharmacokinetic-Evaluable Population

The PK-evaluable population consists of all enrolled participants who received at least 1 dose of itacitinib and provided at least 1 postdose PK sample.

### 6. BASELINE, EXPOSURE, AND DISPOSITION

Appendix A provides a list of data displays. Sample data displays are included in a separate document.

### 6.1. Demographics, Baseline Characteristics, and Medical History

Demographics, baseline characteristics, medical history, lung transplant history, BOS history, prior and concomitant medications for immunosuppression, and prior and concomitant medications for treatment of BOS will be summarized for the FAS and listed. Procedures and nondrug therapies will be listed for the FAS.

### 6.1.1. Demographics and Baseline Characteristics

Demographics and baseline characteristics include the following: age, sex, race, ethnicity, weight, height, and BMI.

### **6.1.2. Medical History**

For participants in the FAS, medical history will be summarized. This summation will include the number and percentage of participants with significant medical history for each body system/organ class as documented on the eCRF.

#### 6.1.3. Lung Transplant History

Time since double lung transplant, indication for transplant, donor CMV status, recipient CMV status, donor EBV status, recipient EBV status, history of acute rejection, history of primary graft dysfunction, history of donor-specific antibodies, history of gastroesophageal reflux disease, history of CMV pneumonitis, history of colonization with aspergillus, post-transplant baseline FEV<sub>1</sub> (absolute and % predicted), and best post-transplant forced vital capacity will be summarized descriptively. Among these variables, summaries for continuous variables will include but not be limited to the number of observations, mean, standard deviation, median, minimum, and maximum. Summaries for categorical variables will include the number and percentage of participants in each category.

#### 6.1.4. Bronchiolitis Obliterans Syndrome History

Time since BOS diagnosis, BOS grade at diagnosis, BOS grade at screening, augmented immunosuppression since onset of BOS (other than ECP), and ECP will be summarized.

### **6.1.5.** Medications for Immunosuppression

Medications for immunosuppression will be coded using the WHO Drug Dictionary. For participants in the FAS, the number and percentage of participants with medications for immunosuppression will be summarized separately for the 3 categories of induction, maintenance, and treatment for acute rejection. Within each category, the summary will be by WHO drug class and WHO drug term.

#### 6.1.6. Medications for Treatment of Bronchiolitis Obliterans Syndrome

Prior medications for treatment of BOS will be coded using the WHO Drug Dictionary. For participants in the FAS, the number and percentage of participants with prior medications for treatment of BOS will be summarized by WHO drug class and WHO drug term.

### **6.2.** Disposition of Participants

The number and percentage of participants who were randomized, who were treated, who discontinued study treatment with a primary reason for discontinuation, and who withdrew from the study with a primary reason for withdrawal will be summarized for the FAS. The number of participants enrolled by country and/or site will also be provided by treatment group.

#### **6.3.** Protocol Deviations

Protocol deviations recorded on the eCRF will be summarized and listed.

### 6.4. Exposure

For participants in the FAS, exposure to itacitinib will be summarized descriptively as follows:

#### • Duration of treatment with itacitinib:

Duration of treatment (days) = date of last dose of itacitinib – date of first dose of itacitinib + 1

### • Average daily dose of itacitinib:

Average daily dose of itacitinib (mg/day) = [total actual dose taken (mg)] / [duration of treatment with itacitinib (days) – days of itacitinib interruption]

#### • Dose modifications of itacitinib:

Number of participants who had itacitinib dose reduction and/or interruption

# 6.5. Study Drug Compliance

For participants in the FAS, overall compliance (%) for itacitinib will be calculated for all participants as follows:

Overall compliance (%) =  $100 \times [\text{total dose actually taken (mg)}] / [\text{total prescribed dose (mg)}]$ 

The total prescribed dose is defined as the sum of the doses prescribed by the investigator accounting for dose modifications.

#### 6.6. Prior and Concomitant Medication

Prior medications and concomitant medications (excluding medications for immunosuppression and treatment for BOS) will be coded using the WHO Drug Dictionary. For participants in the FAS, the number and percentage of participants each with prior and concomitant medications will be summarized by WHO drug class and WHO drug term. In the data listing, each medication will be recorded as prior, concomitant, or both prior and concomitant.

#### 7. EFFICACY

Appendix A provides a list of data displays. Sample data displays are included in a separate document.

### 7.1. General Considerations

All efficacy analyses will be done by treatment group using the FAS. The SGRQ Total Score, QOL-SF-12 Questionnaire, and EQ-5D-3L analyses will not be performed due to the early study termination.

For continuous measurements, summary statistics will include sample size, mean, median, standard deviation, standard error of the mean, minimum, and maximum. For all continuous variables, both the actual value and change and/or percentage from baseline (if available) will be analyzed. For categorical measurements, summary statistics will include sample size, frequency, and percentages.

All by-visit analyses will include the EOT and follow-up visits if the data are available.

### 7.2. Efficacy Hypotheses

Not applicable.

### 7.3. Analysis of the Primary Efficacy Parameter

In Phase 1, the primary endpoint is FEV<sub>1</sub>. Change and percentage change from baseline in FEV<sub>1</sub> and FEV<sub>1</sub> % predicted will be summarized by visit and treatment group.

In Phase 2, the primary endpoint is  $FEV_1$  response rate through the Week 12 visit, defined as the proportion of participants demonstrating a  $\geq 10\%$  absolute increase in  $FEV_1$  compared with baseline, confirmed by 2 consecutive spirometric assessments  $\geq 1$  week apart. The primary analysis will be conducted once the last participant completes the Week 12 visit or withdraws from the study. If a participant withdraws from the study before Week 12, or there is no  $FEV_1$  data up to and including Week 12, the participant will be considered as a nonresponder. Summary statistics and 95% CIs will be provided. Confidence intervals will be calculated based on the exact method for binomial distributions.

In Phase 1,  $FEV_1$  response rate will also be calculated due to the fact that duration of  $FEV_1$  response is a secondary efficacy endpoint in Phase 1.

# 7.4. Analysis of the Secondary Efficacy Parameter

#### 7.4.1. Duration of FEV<sub>1</sub> Response

Duration of FEV<sub>1</sub> response is defined as the interval between the onset of response and the earliest of BOS progression, loss of clinical benefit as determined by the investigator, or death, in which:

• The time of onset of response is defined as the earliest assessment date when ≥ 10% absolute increase in FEV<sub>1</sub> compared with pretreatment baseline (confirmed by 2 consecutive spirometric assessments ≥ 1 week apart) is achieved.

- BOS progression is defined as ≥ 10% absolute decrease in FEV<sub>1</sub> compared with
  pretreatment baseline observed in at least 2 consecutive spirometric assessments at least
  3 weeks apart. The onset of BOS progression is the earliest date of such qualified
  assessments.
- Time of loss of clinical benefit is the date when a participant discontinues treatment due to "lack of efficacy."

Participants with no observed BOS progression, loss of clinical benefit, or death at the time of database lock or discontinuation will be censored at the time of last valid FEV<sub>1</sub> assessment.

Duration of FEV<sub>1</sub> response will be assessed using the Kaplan-Meier method for participants who achieve a response. Median duration and 95% CIs will be estimated.

### 7.4.2. Time to Progression or Death

Time to progression or death, defined as the interval between the start of itacitinib treatment and BOS progression (defined as a  $\geq$  10% absolute decrease in FEV<sub>1</sub> from pretreatment baseline observed in at least 2 consecutive spirometric assessments at least 3 weeks apart) or death. The time of BOS progression follows the same definition as in Section 7.4.1. Participants with no observed BOS progression or death at the time of database lock or discontinuation will be censored at the time of last valid FEV<sub>1</sub> assessment.

Time to progression or death will be estimated by the Kaplan-Meier method. Median duration and 95% CIs will be estimated.

#### 7.4.3. SGRQ Total Score

The SGRQ (Jones et al 1991) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airway disease. It consists of 50 items covering 3 domains: symptoms (8 items), activity (16 items), and impacts (26 items).

A component score will be calculated for each of the 3 domains. If more than 2 items in the symptoms domain are missing, the symptom component score will set to be missing. If more than 4 items in the activity domain are missing, the activity component score will set to be missing. If more than 6 items in the impacts domain are missing, the impacts component score will set to be missing.

One total score will be calculated if none of the component scores is missing. All scales have a score range between 0 and 100 with higher scores indicating a worse quality of life.

Summary statistics will be provided for change from baseline in SGRQ component scores and the total score at each scheduled visit.

#### 7.4.4. QOL-SF-12 Questionnaire

The QOL-SF-12 v2 (Ware et al 1996) is a 12-item subset of the QOL-SF-36 v2 scale that captures changes in health status during the course of treatment. The QOL-SF-12 assesses 8 health concepts related to limitations in physical activities, social activities, bodily pain, general mental and physical health, and vitality.

For this questionnaire, 1 component score will be provided for each of 8 health concepts. Two summary scores, physical component summary and mental component summary, will also be provided. For each item, a higher score indicates a better health state.

Summary statistics will be provided for change from baseline in 2 scales at each scheduled visit.

#### 7.4.5. EQ-5D-3L

The EQ-5D-3L (EuroQol Research Foundation 2017) essentially consists of 2 components: the EQ-5D descriptive scale and the EQ-VAS.

The EQ-5D-3L descriptive system comprises the following 5 dimensions, each describing a different aspect of health: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. Each dimension has 3 levels: no problems, some problems, and extreme problems. The EQ-VAS records the respondent's self-rated health on a vertical visual analog scale on which the endpoints are labeled as "the best health you can imagine" and "the worst health you can imagine."

At each specific visit (starting on Day 1), the participant will be asked to indicate their health state. Missing values will not be imputed. The categorical outcomes for the 5 dimensions (mobility, self-care, usual activities, anxiety/depression, and pain/discomfort) will be summarized by visit, and summary statistics will include frequency and percentage. The change from baseline in EQ-VAS score will be summarized.

#### 8. PHARMACOKINETICS AND PHARMACODYNAMICS

### 8.1. Pharmacokinetic Analyses

#### 8.1.1. Pharmacokinetic Data

Participants will arrive at the clinic having withheld their morning dose of itacitinib. Pharmacokinetic samples will be obtained at the visits indicated in Protocol Table 3. After the predose PK sample is drawn, participants will take the dose of itacitinib. Predose is defined as within 24 hours before administration of itacitinib. The exact date and time of the PK blood draws will be recorded on the eCRF along with the date and time of the last dose of study drug and details of the last meal before the blood draw. Instructions for sample preparation and shipping will be provided in the Laboratory Manual. Sample collection times and windows for itacitinib are shown in Table 2. Adjustments to the timing of blood sampling postdose may be made based on emerging PK data; however, no more than 6 postdose timepoints will be used, and the maximum scheduled timepoint will be no greater than 12 hours postdose.

**Table 2:** Sample Collection Times for Pharmacokinetic Assessments of Itacitinib

| Visit | Timing of Sample Relative to Itacitinib Administration | | | |
|---|---|---|---|---|
| Baseline (Day 1) <sup>a</sup> | Predose | $1 \text{ h} \pm 15 \text{ min}$ | $2 h \pm 30 min$ | 5 h ± 60 min |
| Week 4 | Predose (-30 min) | 1 h ± 15 min | 2 h ± 30 min | 5 h ± 60 min |

<sup>&</sup>lt;sup>a</sup> Phase 1 participants only.

# 8.1.2. Participant Demographic, Clinical Laboratory, Disease-Related, and Pharmacogenomic Variables and Concomitant Medications

Participant demographic assessments (eg, age, weight, BMI, sex, race) and clinical laboratory measurements (eg, FEV<sub>1</sub>, creatinine clearance, serum albumin, total bilirubin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase) may be explored as time-independent predictors of PK variability. Concomitant medications may be explored as time-dependent covariates in the population PK analysis.

#### 8.1.3. Pharmacokinetic Analyses

| The noncompartmental analysis for itacitinib PK will be performed using WinNonlin® v8.0 or later (Certara, Princeton, NJ). The following PK parameters will be estimated where possible: $C_{max}$ , $t_{max}$ , $C_{min}$ , $AUC_{0-t}$ , $AUC_{0-\tau}$ , $t_{1/2}$ , $Cl/F$ , and $V_z/F$ . |
|---|



### **8.1.4.** Report

A PK report will be prepared to include listings of observed itacitinib plasma concentration data and estimated PK parameters in accordance with guidance of both US and EU regulatory authorities.

### 8.2. Pharmacodynamic Analyses

Baseline and pharmacodynamic analyses of serum cytokines, will be conducted as follows:

- Baseline differences in inflammatory mediators between responders and nonresponders will be assessed using:
  - Unadjusted logistic regression models, with FEV<sub>1</sub> response as a binary variable.
  - Unadjusted general linear models, with change in FEV<sub>1</sub> as a continuous variable.
  - Statistically significant unadjusted models will be adjusted for baseline FEV<sub>1</sub>, age, sex, itacitinib dose, and prior immunosuppressive therapy. If fewer than 10 observations are available per covariate, covariates will be removed in order from weakest to strongest statistical association with the inflammatory mediator (outcome) of interest, until at least 10 observations per covariate are available. Alternatively, if variables are determined to be biologically relevant to the analysis, the model will include the principal component analysis scores for the covariates. Only scores with eigenvalues > 1 will be included.
- Pharmacodynamic changes from baseline will be compared between responders and nonresponders using paired t-tests.
- Significance will be reported at p < 0.05 and fold change > |15%|.

#### 9. SAFETY AND TOLERABILITY

Appendix A provides a list of data displays. Sample data displays are included in a separate document.

#### 9.1. General Considerations

All safety analyses will be conducted using the FAS and summarized by treatment group.

#### 9.2. Adverse Events

#### 9.2.1. Adverse Event Definitions

A TEAE is either an AE reported for the first time or worsening of a pre-existing event after first dose of itacitinib until 30 days after the last dose of itacitinib. Analysis of AEs will be limited to TEAEs, but data listings will include all AEs regardless of their timing in relation to the administration of itacitinib.

Adverse events will be tabulated by MedDRA PT and SOC. Severity of AEs will be described and graded using the NCI CTCAE v5.0 (2017). The CTCAE reporting guidelines and grading details are available on the Cancer Therapy Evaluation Program website.

A grading (severity) scale is provided for each AE term. If the toxicity is not included in the CTCAE v5.0 criteria, then it will be rated on a scale of 1 to 4 as follows: 1 = mild, 2 = moderate, 3 = severe, and 4 = life-threatening. All toxicities will be graded based on the worst level reached, not the level they may have reached if they had not been treated. When the intensity of an AE changes over time for a reporting period (eg, between visits), then each change in intensity will be reported as an AE until the event resolves.

The subset of AEs considered by the investigator to be related to itacitinib will be considered to be treatment-related AEs. If the investigator does not specify the relationship of the AE to itacitinib, then the AE will be considered to be treatment-related. The incidence of AEs and treatment-related AEs will be tabulated. Serious AEs will also be tabulated.

Any missing onset date, causality, or severity must be queried for resolution. Unsolved missing values will be handled according to the following rules:

- An unsolved missing causality will be considered treatment-related.
- An unsolved missing severity will be identified as an unknown severity.

For purposes of analysis, all AEs will be considered TEAEs unless the AE can unequivocally be defined as not treatment-emergent.

#### 9.2.2. Adverse Event Summaries

An overall summary of AEs by treatment group will include:

- Number (%) of participants reporting any TEAEs
- Number (%) of participants reporting any serious TEAEs
- Number (%) of participants reporting any Grade 3 or higher TEAEs
- Number (%) of participants reporting any TEAEs related to itacitinib

- Number (%) of participants who temporarily interrupted itacitinib because of TEAEs
- Number (%) of participants with itacitinib dose reduction because of TEAEs
- Number (%) of participants who permanently discontinued itacitinib because of TEAEs
- Number (%) of participants who had a fatal TEAE

The following summaries will be produced by MedDRA term:

- Summary of TEAEs by MedDRA SOC and PT
- Summary of TEAEs by MedDRA PT in decreasing order of frequency
- Summary of TEAEs by MedDRA SOC, PT, and maximum severity
- Summary of Grade 3 or higher TEAEs by MedDRA SOC and PT
- Summary of Grade 3 or higher TEAEs by MedDRA PT in decreasing order of frequency
- Summary of serious TEAEs by MedDRA SOC and PT
- Summary of serious TEAEs by MedDRA PT in decreasing order of frequency
- Summary of itacitinib treatment-related TEAEs by MedDRA SOC and PT
- Summary of itacitinib treatment-related TEAEs by MedDRA PT in decreasing order of frequency
- Summary of itacitinib treatment-related serious TEAEs by MedDRA SOC and PT
- Summary of TEAEs with a fatal outcome by MedDRA SOC and PT
- Summary of TEAEs leading to discontinuation of itacitinib by MedDRA SOC and PT
- Summary of TEAEs leading to itacitinib dose reduction by MedDRA SOC and PT
- Summary of TEAEs leading to itacitinib dose interruption by MedDRA SOC and PT

# 9.2.3. Clinically Notable Treatment-Emergent Adverse Events Based on Customized MedDRA Queries

The following categories of clinically notable events will be summarized based on customized MedDRA queries (see Appendix B):

- Anemia
- Neutropenia
- Thrombocytopenia
- QT prolongation
- Hyperlipidemia
- EBV infection
- CMV infection

Within each category, the number and percentage of participants with at least 1 TEAE occurring during the treatment phase tabulated by MedDRA PT will be summarized. Summaries of clinically notable TEAEs based on customized MedDRA queries will be provided by treatment group, category, PT, and the highest grade or outcome as follows:

- Overall summary of clinically notable TEAEs in the treatment phase based on customized MedDRA queries.
- Number (%) of participants with clinically notable TEAEs in the treatment phase based on customized MedDRA queries by PT and outcome.
- Number (%) of participants with clinically notable TEAEs in the treatment phase based on customized MedDRA queries by PT and highest grade.

### 9.3. Clinical Laboratory Tests

Laboratory values and change from baseline values will be summarized descriptively by visit. Baseline will be determined according to Section 4.1.3. If there are multiple values that meet the criteria for baseline, additional rules may be provided after consultation with the medical monitor to delineate which value will be defined as baseline.

Summaries for abnormally high and abnormally low laboratory values will be provided when the laboratory parameter has both high and low grading criteria.

For test results that will be summarized with available normal ranges, the number and percentage of participants with the laboratory values being low (but never high), normal, high (but never low), and both low and high will be calculated for each test. This shift summary will be produced for each parameter for the FAS. The denominator for the percentage calculation will use the number of participants in the baseline category (ie, low, high, normal, missing) as the denominator for the percentage in each of the categories during the study.

Severity grades will be assigned to laboratory test values based on the numerical component of CTCAE v5. Shift tables will be presented showing change in CTCAE grade from baseline to worst grade postbaseline. The denominator for the percentage calculation will be the number of participants in the baseline category.

# 9.4. Vital Signs

Descriptive statistics and mean change from baseline will be summarized for vital signs (blood pressure, pulse, respiratory rate, and body temperature) at each assessment time by treatment group. Vital sign results will be reviewed for abnormal values (see Table 3), and participants exhibiting abnormal vital sign values will be summarized and listed. A value will be considered an "alert" value if it is outside the established range and shows a > 25% change from baseline. The values for participants exhibiting alert vital sign abnormalities will be summarized and listed.

**Table 3:** Criteria for Vital Sign Abnormalities

| Parameter | High Threshold | Low Threshold |
|--------------------------|------------------|-----------------|
| Systolic blood pressure | > 155 mmHg | < 85 mmHg |
| Diastolic blood pressure | > 100 mmHg | < 40 mmHg |
| Pulse | > 100 bpm | < 45 bpm |
| Temperature | > 38°C | < 35.5°C |
| Respiratory rate | > 24 breaths/min | < 8 breaths/min |

### 9.5. Electrocardiograms

Twelve-lead ECGs including PR, RR, QT, QRS, QTcB, and QTcF intervals will be obtained for each participant during the study. Abnormal ranges for ECG values are defined in Table 4. Electrocardiogram values will also be considered abnormal if the absolute percentage change from baseline is more than 25%. Participants exhibiting ECG abnormalities will be listed with study visit and assigned treatment group. Abnormal values for participant with alert ECG values, defined as both the absolute value and the percentage change from baseline being outside normal ranges, will be identified and listed. Clinically significant ECG values, in the judgment of the investigator, will also be summarized and listed.

**Table 4:** Criteria for Electrocardiogram Abnormalities

| Parameter | High Threshold | Low Threshold |
|-----------|----------------|---------------|
| QTcF/QTcB | > 450 ms | < 295 ms |
| PR | > 220 ms | < 75 ms |
| QRS | > 120 ms | < 50 ms |
| QT | > 500 ms | < 300 ms |
| RR | > 1330 ms | < 600 ms |

#### 10. INTERIM ANALYSES

No formal interim analysis is planned. A steering committee meeting will occur at the end of Phase 1 for RP2D dose determination, for which an informal analysis of safety and efficacy data will be performed.

#### 11. CHANGES AND MODIFICATIONS TO THE ANALYSIS PLAN

All versions of the SAP are listed in Table 5.

**Table 5:** Statistical Analysis Plan Versions

| SAP Version | Date |
|-------------|-------------|
| Original | 12 APR 2023 |
| Amendment 1 | 26 AUG 2024 |

### 11.1. Changes to Protocol-Defined Analyses

Not applicable.

## 11.2. Changes to the Statistical Analysis Plan

#### **11.2.1. Amendment 1**

The following updates were made for SAP Amendment 1 to align with early study termination:

- The planned tables, figures, and listings were updated in Appendix A to remove those that were not needed.
- Analyses for SGRQ Total Score, QOL-SF-12 Questionnaire, and EQ-5D-3L were removed.
- Text was updated to address the analyses not being performed.

Other minor administrative changes have been incorporated throughout and are noted in the redline version of the document.

#### 12. REFERENCES

Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.

EuroQol Research Foundation. EQ-5D-3L. Accessed January 31, 2023.https://euroqol.org/eq-5d-instruments/eq-5d-3l-about/

Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med 1991;85 Suppl B:25-37.

National Cancer Institute. Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. 2017.

Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care 1996;34:220-233.

# APPENDIX A. PLANNED TABLES, FIGURES, AND LISTINGS

This appendix provides a list of the planned tables, figures, and listings. Standard tables will follow the conventions in the Standard Safety Tables current version if necessary.

#### **Tables**

| Table No. | Title | Population |
|---|---|---|
| Baseline and | Baseline and Demographic Characteristics | |
| 1.1.1 | Analysis Populations | All Screened |
| 1.1.2 | Summary of Participant Disposition | FAS |
| 1.1.3 | Summary of Number of Participants Enrolled by Site | FAS |
| 1.1.4 | Summary of Protocol Deviations | FAS |
| 1.2.1 | Summary of Demographics and Baseline Characteristics | FAS |
| Efficacy | | |
| 2.1 | Summary of FEV <sub>1</sub> Response | FAS |
| 2.2.1 | Summary of FEV <sub>1</sub> by Visit | FAS |
| 2.3.1 | Summary of Duration of FEV <sub>1</sub> Response | FAS |
| 2.3.2 | Summary of Time to Progression or Death | FAS |
| Safety | | |
| 3.1.1 | Summary of Exposure and Duration of Exposure to Itacitinib | FAS |
| 3.1.2 | Summary of Study Drug Compliance | FAS |
| 3.2.1 | Overall Summary of Treatment-Emergent Adverse Events | FAS |
| 3.2.2 | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ<br>Class and Preferred Term | FAS |
| 3.2.3 | Summary of Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | FAS |
| 3.2.4 | Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term, and Maximum Severity | FAS |
| 3.2.5 | Summary of Grade 3 or Higher Treatment-Emergent Adverse Events by<br>MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.7 | Summary of Serious Treatment-Emergent Adverse Events by MedDRA<br>System Organ Class and Preferred Term | FAS |
| 3.2.9 | Summary of Itacitinib Treatment-Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.10 | Summary of Itacitinib Treatment-Related Treatment-Emergent Adverse Events by MedDRA Preferred Term in Decreasing Order of Frequency | FAS |
| 3.2.11 | Summary of Itacitinib Treatment-Related Serious Treatment-Emergent<br>Adverse Events by MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.12 | Summary of Treatment-Emergent Adverse Events With a Fatal Outcome by MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.13 | Summary of Treatment-Emergent Adverse Events Leading to Discontinuation of Itacitinib by MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.14 | Summary of Treatment-Emergent Adverse Events Leading to Itacitinib Dose<br>Reduction by MedDRA System Organ Class and Preferred Term | FAS |
| 3.2.15 | Summary of Treatment-Emergent Adverse Events Leading to Itacitinib Dose Interruption by MedDRA System Organ Class and Preferred Term | FAS |

# Listings

| Listing No. | Title |
|---|---|
| Baseline Den | Baseline Demographic and Characteristic |
| 2.1.1 | Participant Enrollment and Disposition Status |
| 2.2.1 | Protocol Deviations |
| 2.4.1 | Demographic and Baseline Characteristics |
| 2.4.2 | Lung Transplant History |
| 2.4.3 | Bronchiolitis Obliterans Syndrome History |
| 2.4.4 | Medications for Immunosuppression |
| 2.4.5 | Medications for Treatment of Bronchiolitis Obliterans Syndrome |
| 2.4.6 | Prior and Concomitant Medications |
| 2.4.7 | Medical History |
| 2.5.1 | Itacitinib Exposure and Compliance |
| Efficacy | Efficacy |
| 2.6.1 | FEV <sub>1</sub> Assessment |
| 2.6.2 | FEV <sub>1</sub> Response Assessment |
| 2.6.3 | Time to Progression or Death Events and Assessment |
| 2.6.4 | Duration of FEV <sub>1</sub> Response Events and Assessment |
| 2.6.6 | Deaths |
| Safety | |
| 2.7.1 | Adverse Events |
| 2.7.2 | Serious Adverse Events |
| 2.7.3 | Grade 3 and Higher Adverse Events |
| 2.7.4 | Fatal Adverse Events |
| 2.7.5 | Treatment-Related Adverse Events |
| 2.7.6 | Adverse Events Leading to Interruption, Reduction, or Discontinuation of Itacitinib |
| 2.8.1 | Clinical Laboratory Values – Hematology |
| 2.8.2 | Clinical Laboratory Values – Chemistry |
| 2.8.3 | Clinical Laboratory Values – Coagulation |
| 2.8.4 | Clinical Laboratory Values – Lipid Panel |
| 2.9.1 | Vital Signs |
| 2.10.1 | 12-Lead ECG |
| 2.10.2 | Abnormal 12-Lead ECG Values |
| 2.10.4 | Clinically Significant 12-Lead ECG Values |

# APPENDIX B. CLINICALLY NOTABLE EVENTS BASED ON CUSTOMIZED MEDDRA QUERIES

This appendix provides the categories of clinically notable events based on customized MedDRA queries.

### **Clinically Notable Hematological Events**

| Category | Preferred Term |
|------------------|-------------------------------------------|
| Anemia | Anaemia macrocytic |
| Anemia | Aplasia pure red cell |
| Anemia | Aplastic anaemia |
| Anemia | Erythroblast count decreased |
| Anemia | Erythropenia |
| Anemia | Hypoplastic anaemia |
| Anemia | Microcytic anaemia |
| Anemia | Red blood cell count decreased |
| Anemia | Anaemia |
| Anemia | Haematocrit decreased |
| Anemia | Haemoglobin decreased |
| Anemia | Leukoerythroblastic anaemia |
| Neutropenia | Agranulocytosis |
| Neutropenia | Band neutrophil count decreased |
| Neutropenia | Febrile neutropenia |
| Neutropenia | Granulocyte count decreased |
| Neutropenia | Granulocytopenia |
| Neutropenia | Neutropenia |
| Neutropenia | Neutropenic infection |
| Neutropenia | Neutropenic sepsis |
| Neutropenia | Neutrophil count decreased |
| Thrombocytopenia | Acquired amegakaryocytic thrombocytopenia |
| Thrombocytopenia | Platelet count decreased |
| Thrombocytopenia | Thrombocytopenia |
| Thrombocytopenia | Plateletcrit decreased |

# **Hematological Infection**

| Category | Preferred Term |
|---|---|
| EBV infection | Epstein-Barr virus positive mucocutaneous ulcer |
| EBV infection | Epstein-Barr viraemia |
| EBV infection | Epstein-Barr virus associated lymphoma |
| EBV infection | Epstein-Barr virus associated lymphoproliferative disorder |
| EBV infection | Epstein-Barr virus infection |
| EBV infection | Hepatitis infectious mononucleosis |
| EBV infection | Infectious mononucleosis |
| EBV infection | Oral hairy leukoplakia |
| EBV infection | Post transplant lymphoproliferative disorder |
| EBV infection | X-linked lymphoproliferative syndrome |
| EBV infection | Epstein-Barr virus test positive |
| EBV infection | Epstein-Barr virus antibody positive |
| Cytomegaloviral infections | Congenital cytomegalovirus infection |
| Cytomegaloviral infections | Cytomegalovirus chorioretinitis |
| Cytomegaloviral infections | Cytomegalovirus colitis |
| Cytomegaloviral infections | Cytomegalovirus duodenitis |
| Cytomegaloviral infections | Cytomegalovirus enteritis |
| Cytomegaloviral infections | Cytomegalovirus enterocolitis |
| Cytomegaloviral infections | Cytomegalovirus gastritis |
| Cytomegaloviral infections | Cytomegalovirus gastroenteritis |
| Cytomegaloviral infections | Cytomegalovirus gastrointestinal infection |
| Cytomegaloviral infections | Cytomegalovirus gastrointestinal ulcer |
| Cytomegaloviral infections | Cytomegalovirus hepatitis |
| Cytomegaloviral infections | Cytomegalovirus infection |
| Cytomegaloviral infections | Cytomegalovirus mononucleosis |
| Cytomegaloviral infections | Cytomegalovirus mucocutaneous ulcer |
| Cytomegaloviral infections | Cytomegalovirus myelomeningoradiculitis |
| Cytomegaloviral infections | Cytomegalovirus myocarditis |
| Cytomegaloviral infections | Cytomegalovirus nephritis |
| Cytomegaloviral infections | Cytomegalovirus oesophagitis |
| Cytomegaloviral infections | Cytomegalovirus pancreatitis |
| Cytomegaloviral infections | Cytomegalovirus pericarditis |
| Cytomegaloviral infections | Cytomegalovirus syndrome |
| Cytomegaloviral infections | Cytomegalovirus urinary tract infection |
| Cytomegaloviral infections | Cytomegalovirus viraemia |
| Cytomegaloviral infections | Encephalitis cytomegalovirus |
| Cytomegaloviral infections | Disseminated cytomegaloviral infection |
| Cytomegaloviral infections | Pneumonia cytomegaloviral |
| Cytomegaloviral infections | Cytomegalovirus test positive |

# Hyperlipidemia

| Hyperlipidemia Acquired lipoatrophic diabetes Hyperlipidemia Acquired mixed hyperlipidaemia Hyperlipidemia Apolipoprotein B/Apolipoprotein A-1 ratio increased Hyperlipidemia Autoimmune hyperlipidaemia Hyperlipidemia Blood cholesterol abnormal Hyperlipidemia Blood cholesterol esterase increased Hyperlipidemia Blood cholesterol increased Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein particles increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased | Category | Preferred Term |
|---|---|---|
| Hyperlipidemia Apolipoprotein B/Apolipoprotein A-1 ratio increased Hyperlipidemia Autoimmune hyperlipidaemia Hyperlipidemia Blood cholesterol abnormal Hyperlipidemia Blood cholesterol esterase increased Hyperlipidemia Blood cholesterol increased Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlolesterolaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Lipida Intermediate density lipoprotein increased Hyperlipidemia Lipida shormal Hyperlipidemia Lipida shormal Hyperlipidemia Lipida shormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Remnant-like lipoprotein increased Hyperlipidemia Remnant-like lipoprotein increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Acquired lipoatrophic diabetes |
| Hyperlipidemia Autoimmune hyperlipidaemia Hyperlipidemia Blood cholesterol abnormal Hyperlipidemia Blood cholesterol increased Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hyperlipidaemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipida increased Hyperlipidemia Lipida increased Hyperlipidemia Lipida increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Remnant-like lipoprotein increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Acquired mixed hyperlipidaemia |
| Hyperlipidemia Blood cholesterol abnormal Hyperlipidemia Blood cholesterol esterase increased Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia Loburbor Loburbor increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipids protein (a) abnormal Hyperlipidemia Lipids moreased Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein nicreased Hyperlipidemia Remnant-like lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Apolipoprotein B/Apolipoprotein A-1 ratio increased |
| Hyperlipidemia Blood cholesterol esterase increased Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia Hyperlipidemia Hypercholesterolaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Internediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Remnant-like lipoprotein increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Autoimmune hyperlipidaemia |
| Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Libur atto increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein cholesterol increased Hyperlipidemia Low density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Blood cholesterol abnormal |
| Hyperlipidemia Blood triglycerides abnormal Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hyperlipidaemia Hyperlipidemia Lipot natio increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein (a) banormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Remnant-like lipoprotein increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Blood cholesterol esterase increased |
| Hyperlipidemia Blood triglycerides increased Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein cholesterol increased Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Blood cholesterol increased |
| Hyperlipidemia Diabetic dyslipidaemia Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Remnant-like lipoprotein cholesterol increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Blood triglycerides abnormal |
| Hyperlipidemia Dyslipidaemia Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hypercholesterolaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased | Hyperlipidemia | Blood triglycerides increased |
| Hyperlipidemia High density lipoprotein abnormal Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Diabetic dyslipidaemia |
| Hyperlipidemia High density lipoprotein decreased Hyperlipidemia Hypercholesterolaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hypo HDL cholesterolaemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Dyslipidaemia |
| Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia Lipids abnormal Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | High density lipoprotein abnormal |
| Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidaemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia LDL/HDL ratio increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | High density lipoprotein decreased |
| Hyperlipidemia Hypertriglyceridaemia Hyperlipidemia Hypo HDL cholesterolaemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia LDL/HDL ratio increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Remnant-like lipoprotein cholesterol increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Hypercholesterolaemia |
| Hyperlipidemia Hypo HDL cholesterolaemia Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia LDL/HDL ratio increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Hyperlipidaemia |
| Hyperlipidemia Intermediate density lipoprotein increased Hyperlipidemia LDL/HDL ratio increased Hyperlipidemia Lipids abnormal Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Hypertriglyceridaemia |
| Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Hypo HDL cholesterolaemia |
| Hyperlipidemia Lipids abnormal Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Intermediate density lipoprotein increased |
| Hyperlipidemia Lipids increased Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | LDL/HDL ratio increased |
| Hyperlipidemia Lipoprotein (a) abnormal Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipids abnormal |
| Hyperlipidemia Lipoprotein (a) increased Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipids increased |
| Hyperlipidemia Lipoprotein abnormal Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipoprotein (a) abnormal |
| Hyperlipidemia Lipoprotein increased Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipoprotein (a) increased |
| Hyperlipidemia Low density lipoprotein abnormal Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipoprotein abnormal |
| Hyperlipidemia Low density lipoprotein increased Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Lipoprotein increased |
| Hyperlipidemia Non-high-density lipoprotein cholesterol increased Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Low density lipoprotein abnormal |
| Hyperlipidemia Remnant-like lipoprotein particles increased Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Low density lipoprotein increased |
| Hyperlipidemia Total cholesterol/HDL ratio abnormal Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Non-high-density lipoprotein cholesterol increased |
| Hyperlipidemia Total cholesterol/HDL ratio increased Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Remnant-like lipoprotein particles increased |
| Hyperlipidemia Very low density lipoprotein abnormal | Hyperlipidemia | Total cholesterol/HDL ratio abnormal |
| | Hyperlipidemia | Total cholesterol/HDL ratio increased |
| Hyperlipidemia Very low density lipoprotein increased | Hyperlipidemia | Very low density lipoprotein abnormal |
| | Hyperlipidemia | Very low density lipoprotein increased |

# **QT Prolongation**

| Category | Preferred Term |
|-----------------|----------------------------------------|
| QT prolongation | Electrocardiogram QT interval abnormal |
| QT prolongation | Electrocardiogram QT prolonged |
| QT prolongation | Long QT syndrome |
| QT prolongation | Long QT syndrome congenital |
| QT prolongation | Torsade de pointes |
| QT prolongation | Ventricular tachycardia |